CLINICAL TRIAL: NCT03306108
Title: Correlation Between the Neural Response Telemetry (NRT) and Radiological Measurements in Detection of Position of the Electrode Inside the Cochlea
Brief Title: Correlation Between NRT and Radiological Measurements in Detection of Position of the Electrode Inside the Cochlea.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, samah hamdy saeed, principal investigator, Assiut University
Other Study IDs: NRT in Cochlear implantation
Record Dates: First submitted 2017-09-08; First posted 2017-10-10 (Actual); Last update posted 2017-10-10 (Actual); Status verified 2017-09

CONDITIONS: Cochlear Function Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: NRT — NRTratio is based on each individual electrode's ECAP threshold and can identify the intracochlear electrode array position in perimodiolar electrodes. The NRT-ratio showed a good reliability for the determination of the intracochlear electrode array position compared to the radiologic control intraoperatively Calculation of the NRT-ratio is done by dividing the arithmetic average of the t-NRT values from the apical electrodes 16 to 18 divided by the arithmetic average of the basal t-NRT from electrodes 5 to 7. With a NRT-ratio above 1.05, a high chance of a scalar change was rather likely, and a NRT-ratio below 1.05 was associated with a high chance of an electrode array position within the scala tympani.

SUMMARY:
The study will be conducted as Prospective study including 50 patients (aged <6years ) at Otorhinolaryngology department, Assuit University Hospital (aged <6years ) who will undergo cochlear implantation. All subjects will undergo implantation with Medel sonata flex 28 or standard electrodes with a standard surgical procedure. The standard surgical procedure will include extended end aural approach ,posterior tympanotomy and a round window insertion.The results of immediate postoperative Neural Response Telemetry (NRT) measurements & postoperative CT imaging will be obtained.

Each patient will be subjected to the following scheme:

* immediate postoperative Neural Response Telemetry (NRT) measurements
* postoperative CT imaging
* Data obtained from both measurements will be used to determine the intra cochlear electrode position then both data will be correlated.

DETAILED DESCRIPTION:
Cochlear implantation (CI) is a worldwide accepted and effective surgical procedure for patients with profound sensory neural hearing loss to gain near normal hearing.1 The position of electrode inside the cochlea affects the outcomes. Full insertion of the CI electrode array and insertion in scala tympani usually has optimal results and better words recognition.2 Translocation of electrode array from scala tympani to scala vestibule or outword migration of electrode array may result in poor response.2 There are many intraoperative and post operative techniques to determine the position of electrode array inside the cochlea, some are radiological as transorbital view plan x-ray or computed tomography or 3D rotational x ray and others are electrophysiological measurements.3 Although the accuracy of the radiological techinques they are time and cost consuming1. The electrically evoked cochlear action potential (ECAP) threshold is dependent on the distance between the electrodes and the spiral ganglion cells. The neural response telemetry-ratio (NRT-ratio) is one of the electrophysiological measurments techniques and it is based on each individual electrode's ECAP threshold and can identify the intracochlear electrode array position 4. According to a study done by Philipp Mittmann in 2015, a NRT-ratio above 1.05 indicates an electrode translocation from scala tympani to scala vestibuli and a NRT-ratio below 1.05 shows correlation to a pure scala tympani placement5, but another study found variation of the NRT-ratio in a group of patients with an electrode placement within scala tympani.6

ELIGIBILITY:
Inclusion Criteria:

* patients aged < 6years who will undergo cochlear implantation

Exclusion Criteria:

* Revision cochlear implantation.
* incomplete post-operative electrophysiological measurements.
* unfit patients for surgery

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will be conducted as Prospective study at Otorhinolaryngology department, Assuit University Hospital .. All subjects will undergo implantation with Medel sonata flex 28 or standard electrodes with a standard surgical procedure. which will include extended end aural approach ,posterior tympanotomy and a round window insertion.The results of immediate postoperative NRT measurements & postoperative CT imaging will be obtained.
  Each patient will be subjected to the following scheme:
  * immediate postoperative NRT measurements
  * postoperative CT imaging
  * Data obtained from both measurements will be used to determine the intra cochlear electrode position then both data will be correlated.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-10-30 (Estimated); Primary Completion 2018-10 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Value of Neural Response Telemetry (NRT) & Radiological measurments in evaluation of cochlear implant electrode positions | Baseline
  The study will be conducted as Prospective study including 50 patients (aged <6years ) at Otorhinolaryngology department, Assuit University Hospital (aged <6years ) who will undergo cochlear implantation. All subjects will undergo implantation with Medel sonata flex 28 or standard electrodes with a standard surgical procedure. The standard surgical procedure will include extended end aural approach ,posterior tympanotomy and a round window insertion.The results of immediate postoperative Neural Response Telemetry (NRT) measurements & postoperative CT imaging will be obtained.
  Each patient will be subjected to the following scheme:
  * immediate postoperative Neural Response Telemetry (NRT) measurements
  * postoperative CT imaging
  * Data obtained from both measurements will be used to determine the intra cochlear electrode position then both data will be correlated.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Abd El - Aziz, Prof, Study Director
Locations (1):
- Assiut University Hospital, Asyut, Egypt

REFERENCES:
- [Background] Mittmann P, Todt I, Ernst A, Rademacher G, Mutze S, Goricke S, Schlamann M, Lang S, Arweiler-Harbeck D, Christov F. Radiological and NRT-Ratio-Based Estimation of Slim Straight Cochlear Implant Electrode Positions: A Multicenter Study. Ann Otol Rhinol Laryngol. 2017 Jan;126(1):73-78. doi: 10.1177/0003489416675355. Epub 2016 Oct 25. PMID 27780910
- [Background] Mittmann P, Todt I, Ernst A, Rademacher G, Mutze S, Goricke S, Schlamann M, Ramalingam R, Lang S, Christov F, Arweiler-Harbeck D. Electrophysiological detection of scalar changing perimodiolar cochlear electrode arrays: a long term follow-up study. Eur Arch Otorhinolaryngol. 2016 Dec;273(12):4251-4256. doi: 10.1007/s00405-016-4175-2. Epub 2016 Jun 28. PMID 27351885
- [Background] Lathuilliere M, Merklen F, Piron JP, Sicard M, Villemus F, Menjot de Champfleur N, Venail F, Uziel A, Mondain M. Cone-beam computed tomography in children with cochlear implants: The effect of electrode array position on ECAP. Int J Pediatr Otorhinolaryngol. 2017 Jan;92:27-31. doi: 10.1016/j.ijporl.2016.10.033. Epub 2016 Oct 31. PMID 28012529